CLINICAL TRIAL: NCT04233502
Title: A Randomized, Placebo Controlled Study to Investigate the Efficacy and Safety of Slenyto® to Alleviate Sleep Disturbances in Children With Autism Spectrum Disorder
Brief Title: Efficacy and Safety of Slenyto for Insomnia in Children With ASD
Acronym: ASD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was not initiated it was decided to cancel this study
Sponsor: Neurim Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEU_CH_7913
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2020-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental): Slenyto® 1 mg / 5 mg prolonged release Melatonin tablets (pink and yellow) film coated 3 mm in diameter,
  Interventions: Drug: Melatonin
- Placebo melatonin (Placebo Comparator): Placebo melatonin will be identical in appearance (pink and yellow) and formulation to active Slenyto® tablets, but will contain no active melatonin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — prolonged release 1 mg and 5 mg mini-tablets coated odorless and tasteless to facilitate swallowing
  Other Names: Slenyto
  Arms: Melatonin
Drug: Placebo — Placebo melatonin
  Arms: Placebo melatonin

SUMMARY:
This is a randomized placebo controlled study in children diagnosed with autism spectrum disorder (ASD), to Investigate the Efficacy and Safety of Slenyto® to alleviate Sleep Disturbances in these children. .

The main objective is to compare treatment effect of Slenyto® 2 mg or 5 mg to that of placebo on sleep duration (total sleep time [TST]) as assessed by the Sleep and Nap Diary after 3 weeks of double blind treatment.

DETAILED DESCRIPTION:
This is a randomized placebo controlled study in children diagnosed with autism spectrum disorder (ASD). Children will have a documented history of this disorder, as confirmed or consistent with the International Classification of Diseases (ICD 10) or Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (Text Revision; DSM 5) criteria, having DSM-5 criteria based sleep disturbances at screening.

The children will undergo 4 weeks of basic sleep hygiene and behavioral intervention, which will serve as a wash out period from any hypnotics and prohibited medications; Children with a documented history of sleep hygiene and behavioral intervention who are taking a prohibited medication will not require additional training and will undergo a 2-week wash out period before Visit 1.

Children who are still found to be eligible for the study after the 4 week, basic sleep hygiene and behavioral intervention wash out period, will continue in a 2 week single blind (SB) placebo run in period.

. After the 2 week SB placebo run in period (Visit 2; Week 2), children who are still found eligible for study participation will be randomized in a 1:1 ratio to receive either Slenyto® (1 or 5 mg prolonged release melatonin tablets) or placebo for 3 weeks double-blind treatment period. The starting dose will be 2X1mg Slenyto® or matching placebo. During these 3 weeks parents will complete the electronic sleep and nap diary every morning.

After one week of double-blind treatment, on the last day of Week 3 ±3 days (Visit 3), sleep variables will be assessed to determine if dose modification (increase to 1X5 mg Slenyto® or matching placebo) is required. Children will then continue on 2 or 5 mg of Slenyto® or matching placebo to the end of the double blind period (End-of Study Visit 4; Week 5).

Study duration will be either 5, 7, or 9 weeks, including the optional 2-weeks medication wash out and 4 weeks sleep hygiene and behavioral intervention periods (overlapping).

The main objective is to compare treatment effect of Slenyto® 2 mg or 5 mg to that of placebo on sleep duration (total sleep time [TST]) as assessed by the Sleep and Nap Diary after 3 weeks of double blind treatment.

The key secondary endpoints are SL and LSE. Safety will also be assessed by Adverse events, vital signs and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* children 2 to 17.5 years of age at Visit 2 who comply with taking the study drug
* Written informed consent provided by a legal guardian and assent (if needed)
* A documented history of ASD according to or consistent with the ICD 10 or DSM 5 criteria, as confirmed by case note review showing that diagnosis was reached through assessment by a community pediatrician or pediatric neurologist or other health care professionals experienced in the diagnosis who took into account early developmental history and school records.
* Current sleep problems consistent with DSM-5 criteria including: a minimum of 3 months of impaired sleep defined as ≤6 hours of continuous sleep AND ≥ 0.5-hour sleep latency from light off in 3 out of 5 nights based on parent reports and subject medical history. (The maintenance and latency problems do not necessarily have to be in the same 3 nights of the week.)
* May be on a stable dose of non excluded medication for 3 months, including anti epileptics, anti depressants (selective serotonin reuptake inhibitor [SSRIs]), and β blockers. (Only morning administration of β blockers is allowed since β blockers at night have the potential to reduce endogenous
* The sleep disturbance is not due to the direct physiological effects of any concomitant medications such as SSRIs, β blockers etc.

Exclusion Criteria:

* Have had treatment with any form of melatonin within 2 weeks prior to Visit
* Have a known allergy to melatonin or lactose
* Have a known moderate to severe sleep apnea
* Have an untreated medical/ineffectively treated/psychological condition that may be the etiology of sleep disturbances
* Are taking or have been taking prohibited medication within 2 weeks prior to Visit 1
* Are females of child bearing potential that are not using contraceptives and/or breastfeeding and that are sexually active (Abstinence is an acceptable method of contraception.)
* Pregnant females
* Are currently participating in a clinical trial or have participated in a clinical trial involving medicinal product within the last 3 months prior to the study
* Participated in Study NEU_CH_7911
* Children with known renal or hepatic insufficiency

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Total Sleep Time (TST) | after the 3 weeks (Week 5) of double blind treatment
  the change from baseline in average TST time as assessed by a Sleep and Nap Diary

SECONDARY OUTCOMES:
Sleep Latency (SL) | after 3 weeks (Week 5) of double blind treatment
  • Change from baseline in average SL as assessed by a Sleep and Nap Diary
Longest Sleep Episode (LSE) | after 3 weeks (Week 5) of double blind treatment
  • Change from baseline in average LSE from the Sleep and Nap Diary .

IPD SHARING:
Plan to Share IPD: Undecided